CLINICAL TRIAL: NCT06487572
Title: A Phase 1, Open-label Study to Assess PK Exposures Following Intravenous and Subcutaneous Administration of Risankizumab in Healthy Subjects
Brief Title: A Study to Assess Pharmacokinetic Exposures Following Intravenous and Subcutaneous Administration of Risankizumab in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M24-460
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Risankizumab; ABBV-066
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Risankizumab Dose A for Intravenous (IV) Infusion (Experimental): Participants will receive IV infusion of risankizumab at dose A and then followed for 140 days.
  Interventions: Drug: Risankizumab
- Risankizumab Dose B for Subcutaneous (SC) Injection (Experimental): Participants will receive SC injections of risankizumab at dose B and then followed for 140 days.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Intravenous (IV) Infusion
  Other Names: ABBV-066; SKYRIZI
  Arms: Risankizumab Dose A for Intravenous (IV) Infusion
Drug: Risankizumab — Subcutaneous (SC) Injection
  Other Names: ABBV-066; SKYRIZI
  Arms: Risankizumab Dose B for Subcutaneous (SC) Injection

SUMMARY:
The objective of this study is to compare pharmacokinetic exposures following intravenous and subcutaneous administration of Risankizumab.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 18.0 to ≤ 32.0 kg/m^2 after rounding to the tenths decimal at the time of screening and upon initial confinement. BMI is calculated as weight in kg divided by the square of height measured in meters.
* Body weight greater than 40 kg and less than 100 kg at screening and upon initial confinement.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead ECG

Exclusion Criteria:

* Previous exposure to any anti-interleukin-12/23 or anti interleukin-23 treatment for at least one year prior to Screening.
* Intention to perform strenuous exercise to which the particpant is unaccustomed within one week prior to administration of first dose of study drug and during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to approximately 140 days
  An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Serum Concentration (Cmax) of Risankizumab | Up to approximately 140 days
  Cmax of Risankizumab.
Time to Cmax (Tmax) of Risankizumab | Up to approximately 140 days
  Tmax of Risankizumab.
Area Under the Serum Concentration-Time Curve (AUC) of Risankizumab | Up to approximately Week 4
  AUCt of Risankizumab.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - Clinical Pharmacology Of Miami /ID# 268219, Miami, Florida
  - Acpru /Id# 267057, Grayslake, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-460